CLINICAL TRIAL: NCT03765346
Title: A Single-site, Randomized, Double-blind, Double-dummy, Active-comparator, Placebo-controlled, 3-way Crossover Trial in Adult Non-dependent Recreational Opioid Users to Compare the Intranasal Abuse Potential of Immediate Release Abuse-deterrent and Standard Formulations of Oxycodone
Brief Title: A Comparison of How Likely it is That Different Tablets of Oxycodone Will be Broken up and Snorted by Adults Who Sometimes Take Drugs for Pleasure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HP7030-03; U1111-1203-4920 (Registry Identifier: World Health Organization)
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Substance Abuse
Keywords: intranasal abuse; abuse-deterrent
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxycodone IR ADF and placebo to match oxycodone API (Experimental): Participants receive a single intranasal dose of placebo to match oxycodone API powder (mass of 30 mg) followed by a single intranasal dose of manipulated oxycodone IR ADF (mass of 540 mg, containing oxycodone hydrochloride 30 mg).
  Interventions: Drug: Oxycodone IR ADF; Drug: Placebo to match oxycodone API powder
- Oxycodone API and placebo to match oxycodone IR ADF (Active Comparator): Participants receive a single intranasal dose of oxycodone API powder (mass of 30 mg, containing oxycodone hydrochloride 30 mg) followed by a single intranasal dose of placebo to match manipulated oxycodone IR ADF (mass of 540 mg).
  Interventions: Drug: Oxycodone API powder; Drug: Placebo to match manipulated oxycodone IR ADF.
- Placebo to match oxycodone API and to match oxycodone IR ADF (Placebo Comparator): Participants receive a single intranasal dose of placebo to match oxycodone API powder (mass of 30 mg) followed by a single intranasal dose of placebo to match manipulated oxycodone IR ADF (mass of 540 mg).
  Interventions: Drug: Placebo to match oxycodone API powder; Drug: Placebo to match manipulated oxycodone IR ADF.

INTERVENTIONS:
Drug: Oxycodone IR ADF — Oxycodone IR ADF manipulated/crushed (mass of 540 mg, containing oxycodone hydrochloride 30 mg), in a standardized procedure.
  Arms: Oxycodone IR ADF and placebo to match oxycodone API
Drug: Oxycodone API powder — Oxycodone API powder (mass of 30 mg), containing oxycodone hydrochloride 30 mg.
  Arms: Oxycodone API and placebo to match oxycodone IR ADF
Drug: Placebo to match oxycodone API powder — Placebo to match oxycodone API powder (mass of 30 mg).
  Arms: Oxycodone IR ADF and placebo to match oxycodone API; Placebo to match oxycodone API and to match oxycodone IR ADF
Drug: Placebo to match manipulated oxycodone IR ADF. — Placebo to match oxycodone IR ADF, manipulated (mass of 540 mg).
  Arms: Oxycodone API and placebo to match oxycodone IR ADF; Placebo to match oxycodone API and to match oxycodone IR ADF

SUMMARY:
The trial comprises an Enrollment Visit, a Qualification Phase, a Treatment Phase (including 3 treatment periods), a Final Examination, and a Follow-up Phone Call.

The Qualification Phase includes a naloxone challenge test (to verify that participants are not opioid-dependent) and a drug discrimination test (to determine whether or not participants are able to distinguish intranasally administered active drug from placebo). Participants will be randomized to receive a single intranasal dose each of oxycodone active pharmaceutical ingredient (API) and matching placebo in a double-blind manner. The total mass of each single dose will be 30 milligrams.

Participants who successfully complete the Qualification Phase are eligible to be included in the Treatment Phase. During the Treatment Phase, participants will receive test product, comparator, and placebo following a randomized, double-blind, double-dummy, 3-way crossover design. Participants will receive a single intranasal dose of each of the treatments (combined doses of investigational medicinal product {IMP}) on Day 1, Day 4, and Day 7 of the Treatment Phase. A single dose of a treatment is defined as insufflation of single doses of the 2 applicable IMPs in quick succession. The 2 applicable IMPs must be insufflated in the following pre-defined order. Oxycodone API or placebo to match oxycodone API must always be insufflated first. Oxycodone immediate release (IR) abuse-deterrent formulation (ADF) or placebo to match oxycodone IR ADF must always be insufflated second. The total mass of each single dose of treatment will be 570 milligrams.

ELIGIBILITY:
Inclusion Criteria:

* Participants have given written informed consent to participate.
* Female or male participants, aged 18 years to 55 years inclusive at the time of the Enrollment Visit.
* Body mass index between 20 kilograms per square meter and 32 kilograms per square meter inclusive, with a minimum body weight of 55 kilograms.
* Participants must be in good health as determined by the medical history, physical and laboratory examinations and must not show any clinically significant findings as determined by 12-lead electrocardiogram (ECG), vital signs (pulse rate, respiratory rate, systolic and diastolic blood pressure), oxygen saturation, body temperature, and safety laboratory parameters (hematology, clinical chemistry, clotting, and urinalysis).
* Female participants of childbearing potential must agree to use one of the acceptable contraceptive regimens listed below from at least 15 days prior to the first administration of IMP until at least 30 days after the last administration of IMP.

For female participants of childbearing potential:

* Combined (estrogen- and progestogen-containing) hormonal contraception.
* Progestogen-only hormonal contraception associated with inhibition of ovulation.
* An intra-uterine device (hormone-free).
* An intra-uterine hormone releasing system.
* Bilateral tubal occlusion.
* Double barrier methods (i.e., male condom in addition to diaphragm, spermicide, or contraceptive sponge).

All female participants are considered to be of childbearing potential unless they have undergone hysterectomy or bilateral oophorectomy or have been postmenopausal for at least 12 months (i.e., spontaneous amenorrhea at least 1 year prior to screening and confirmed follicle-stimulating hormone [FSH] level above 40 international units per liter).

* Current opioid users who have used opioids for recreational (non-therapeutic) purposes, i.e., for psychoactive effects, at least 10 times in their lifetime and at least once in the last 12 weeks before the Enrollment Visit.
* Participants who have intranasally insufflated drugs for recreational (non-therapeutic) purposes at least 3 times in the last 12 months before the Enrollment Visit.

Exclusion Criteria:

* Resting pulse rate below 50 beats per minute or above 100 beats per minute.
* Resting systolic blood pressure below 90 mmHg or above 140 mmHg. Resting diastolic blood pressure above 90 mmHg.
* Prolongation of the corrected QT interval (Fridericia), i.e., QTcF above 450 milliseconds, or presence of other of risk factors for torsade de pointes (e.g., heart failure, hypokalemia).
* Evidence for thyroid disease based on clinical and safety laboratory findings, including thyroid-stimulating hormone (TSH).
* Any laboratory value (from blood samples taken at the Enrollment Visit) meeting the following criteria:

  * Out-of-reference range value for serum creatinine or clotting parameter prothrombin international normalized ratio.
  * Exclusion range met for urinalysis or alanine transaminase, aspartate transaminase, alkaline phosphatase, total bilirubin, glucose (fasted), gamma-glutamyl transferase, lactate dehydrogenase, potassium, total protein, sodium, calcium, hemoglobin, hematocrit, white blood cell count, or platelets.
  * Out-of-reference range value for any other safety laboratory parameter that is judged by the investigator to be clinically relevant.
* Positive or missing virus serology test for human immunodeficiency virus Type 1 or Type 2 antibodies and antigen, hepatitis B surface antigen, hepatitis B core antigen antibodies, or hepatitis C virus antibodies.
* For female participants: positive or missing pregnancy test.
* Participant received an IMP or an investigational medical device in another clinical trial less than 30 days before the Enrollment Visit. Depending on the nature of the previous IMP or investigational medical device, a longer washout may be needed.
* Diseases or conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of orthostatic hypotension.
* Known history of or at risk of seizures (i.e., head trauma, epilepsy in family history, unclear loss of consciousness).
* Definite or suspected hypersensitivity to the active substance or to any of the excipients of the IMP; especially known hypersensitivity/intolerance or contraindications to opioids (including [history of] bronchial asthma, chronic obstructive pulmonary disease, pulmonary heart disease, diseases of the adrenal gland, paralytic ileus, prostatic hypertrophy, or urethral stricture), opioid antagonists, or any excipients of the drug formulation.
* Any hint of chronic drug abuse, e.g., injection site (not related to trial procedures).
* Unable to abstain from regular use of any medication (including prescription drugs, over-the-counter drugs, dietary supplements, and herbal remedies like St. John's Wort) from 2 weeks before the Enrollment Visit and anticipated use during the course of the trial. Exempt from this criterion are oral contraceptives in women of childbearing potential and topical medications without systemic effect (except those for intranasal use and nasal sprays).
* Lactating or breastfeeding women.
* Habitually smoking more than 20 cigarettes, 2 cigars, or 2 pipes of tobacco per day in the last 3 months before enrollment in this trial.
* Unable to refrain from smoking or unable to abstain from the use of prohibited nicotine-containing products (including electronic cigarettes, pipes, cigars, chewing tobacco, nicotine topical patches, nicotine gum, or nicotine lozenges) from 1 hour before until 5 hours after each IMP administration.
* Not willing or able to abstain from consumption of beverages or food containing quinine (bitter lemon, tonic water), grapefruit juice (sweet or sour), Seville oranges, or alcohol in the Qualification Phase and the Treatment Phase from 72 hours before the planned first administration of IMP in that phase until discharge from the trial site at the end of that phase.
* Known or suspected of not being able to comply with the requirements of the trial protocol or the instructions of the trial site staff.
* Not able to communicate meaningfully with the trial site staff.
* Employee of the investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial site, as well as family members of the employees or the investigator.
* Blood loss of 500 milliliters or more (e.g., owing to blood donation) less than 56 days before enrollment in this trial.
* Unable to establish reliable venous access.
* Substance or alcohol dependence (excluding nicotine and caffeine) in the last 12 months before enrollment in this trial, as defined by the diagnostic and statistical manual of mental disorders - fourth edition - text revision (DSM-IV-TR).
* Participant has ever participated in or plans to participate in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence.
* Unwillingness or inability to abstain from recreational drug use for the duration of the trial.
* Serious psychiatric or neurological conditions.
* Nasal conditions, e.g., perforated nasal septum, irritated nasal mucosa, obstructed naris.
* History or current evidence of suicidal ideation or suicidal behavior, as assessed by the Columbia-suicide severity rating scale (C-SSRS) ("baseline/screening" version).

Exclusion criteria on Day -1 of the Qualification Phase

* Participation in another clinical trial with an IMP or investigational medical device since enrollment.
* Out-of-reference blood pressure or pulse rate if technical failure can be excluded and result is confirmed by at least 1 additional measurement: systolic blood pressure below 90 mmHg or above 140 mmHg, diastolic blood pressure above 90 mmHg, pulse rate below 50 beats/minute or above 100 beats/minute.
* Withdrawal of informed consent.
* Use of forbidden medication since enrollment in this trial, subject to individual decision by the investigator after consultation with the sponsor.
* Any relevant deterioration in the health of the participant since the Enrollment Visit possibly impacting participation in the trial, at the discretion of the investigator, including: adverse events; vital signs; physical examination, 12-lead ECG (relevant QTcF prolongation, i.e., QTcF above 450 milliseconds); other safety parameters.
* Blood loss of 100 milliliters or more since enrollment in this trial (excluding blood taken for this trial).
* For female participants: positive or missing pregnancy test.
* Positive or missing alcohol test or urine test for drugs of abuse (except for cannabinoids).
* Any hint, especially intravenous or intranasal, of chronic drug abuse, e.g., injection site (not related to trial procedures).
* Failure to comply with trial requirements (e.g., consumption of alcohol, beverages or food containing quinine, grapefruit juice, Seville oranges) judged by the investigator to affect participant safety or interfere with the integrity of the trial.
* Nasal conditions, e.g., perforated nasal septum, irritated nasal mucosa, obstructed naris.
* Current evidence of suicidal ideation or suicidal behavior, as assessed by the C-SSRS ("since last visit" version).
* Clinical opioid withdrawal scale (COWS) score greater than or equal to 5 after administration of naloxone on Day -1 of the Qualification Phase.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Peak effect (Emax) for Drug Liking "at this moment". | at 0.16, 0.33, 0.5, 0.75, 1, 1.33, 1.66, 2, 3, 4, 6, 8, 10, 12 hours, and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  100-point bipolar visual analog scale (VAS) ratings after each IMP administration in response to the statement "At this moment, my liking for this drug is". The 100 millimeter (mm) bipolar VAS is anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), to the left with "strong disliking" (score of 0 mm) and to the right with "strong liking" (score of 100 mm).

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of oxycodone | pre-dose and at 0.16, 0.33, 0.5, 0.75, 1, 1.33, 1.66, 2, 3, 4, 6, 8, 10, 12 hours, and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  The analysis in plasma will be performed by means of a validated LC-MS/MS method.
Area under the plasma concentration-time curve of oxycodone from time point 0 to t (AUC0-t) | pre-dose and at 0.16, 0.33, 0.5, 0.75, 1, 1.33, 1.66, 2, 3, 4, 6, 8, 10, 12 hours, and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  The analysis in plasma will be performed by means of a validated LC-MS/MS method.
Area under the plasma concentration-time curve of oxycodone from time point 0 to infinity (AUC) | pre-dose and at 0.16, 0.33, 0.5, 0.75, 1, 1.33, 1.66, 2, 3, 4, 6, 8, 10, 12 hours, and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  The analysis in plasma will be performed by means of a validated LC-MS/MS method.
High: 100-point unipolar VAS | at 0.16, 0.33, 0.5, 0.75, 1, 1.33, 1.66, 2, 3, 4, 6, 8, 10, 12 hours, and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  100-point unipolar VAS ratings after each IMP administration in response to the statement "At this moment, I am feeling high". The 100 mm unipolar VAS is anchored to the left with "not at all" (score of 0 mm) and to the right with "extremely" (score of 100).
Overall Drug Liking: 100-point bipolar VAS | at 12 and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  100-point bipolar VAS ratings after each IMP administration in response to the statement "Overall, my liking for this drug is". The 100 mm bipolar VAS is anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), to the left with "strong disliking" (score of 0 mm) and to the right with "strong liking" (score of 100 mm).
Take Drug Again: 100-point bipolar VAS | at 12 and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  100-point bipolar VAS ratings after each IMP administration in response to the statement "I would take this drug again". The 100 mm bipolar VAS is anchored in the center with a neutral anchor of "neutral" (score of 50 mm), to the left with "definitely not" (score of 0 mm) and to the right with "definitely so" (score of 100 mm).
Bad Effects: 100-point unipolar VAS | at 0.16, 0.33, 0.5, 0.75, 1, 1.33, 1.66, 2, 3, 4, 6, 8, 10, 12 hours, and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  100-point unipolar VAS ratings after each IMP administration in response to the statement "At this moment, I can feel bad drug effects". The 100 mm unipolar VAS, is anchored to the left with "not at all" (score of 0 mm) and to the right with "extremely" (score of 100).
Ease Of Snorting: 100-point bipolar VAS | at 0 hour as soon as possible after IMP administration on Day 1, Day 4, and Day 7
  100-point bipolar VAS ratings after each IMP administration in response to the statement "How easy was it to snort?". The 100 mm bipolar VAS is anchored in the center with a neutral anchor of "neither easy nor difficult" (score of 50 mm), to the left with "very difficult" (score of 0 mm) and to the right with "very easy" (score of 100 mm).
Pleasantness Of Snorting: 100-point bipolar VAS | at 0 hour as soon as possible after IMP administration on Day 1, Day 4, and Day 7
  100-point bipolar VAS ratings after each IMP administration in response to the statement "How does it feel in your nose?". The 100 mm bipolar VAS is anchored in the center with a neutral anchor of "neither pleasant nor unpleasant" (score of 50 mm), to the left with "very unpleasant" (score of 0 mm) and to the right with "very pleasant" (score of 100 mm).
Pupillometry parameter: Apparent minimum post dose pupil diameter (PCmin) | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12 hours, and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  The size of the participant's pupil will be measured (in mm) using a pupillometer. The same eye for each participant will be used for all measurements throughout the trial. Measurements will be collected under mesopic lighting conditions. PCmin will be calculated
Pupillometry parameter: Time to reach the apparent minimum diameter (PTmin) | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12 hours, and 24 hours post-dose on Day 1 to 2; Day 4 to 5; and Day 7 to 8
  The size of the participant's pupil will be measured (in mm) using a pupillometer. The same eye for each participant will be used for all measurements throughout the trial. Measurements will be collected under mesopic lighting conditions.
Pupillometry parameter: The area over the curve to 1 hour relative to the baseline (PAOC0-1hour) | Baseline up to 1 hour
  The size of the participant's pupil will be measured (in mm) using a pupillometer. The same eye for each participant will be used for all measurements throughout the trial. Measurements will be collected under mesopic lighting conditions.
Pupillometry parameter: The area over the curve to 8 hours relative to the baseline (PAOC0-8hours) | Baseline up to 8 hours
  The size of the participant's pupil will be measured (in mm) using a pupillometer. The same eye for each participant will be used for all measurements throughout the trial. Measurements will be collected under mesopic lighting conditions.
Incidence of adverse events of manipulated IMP | From the first IMP administration (Day 1) to the Final Examination (Day 9)
  Number of adverse events and number of participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Algorithme Pharma, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No